CLINICAL TRIAL: NCT04168086
Title: Dissecting Cerebellar Functions in Visuomotor Adaptation With Transcranial Focused Ultrasound Stimulation
Brief Title: Cerebellar Functions in Visuomotor Adaptation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Virginia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 21135
Record Dates: First submitted 2019-03-19; First posted 2019-11-19 (Actual); Last update posted 2019-11-19 (Actual); Status verified 2019-11

CONDITIONS: Healthy Participants
Keywords: Ultrasound; Neuromodulation; Cerebellum; Transcranial Ultrasound Stimulation
MeSH Terms: interventions — salicylhydroxamic acid

STUDY DESIGN:
Who Masked: Participant
Masking Description: Participants will be blinded to what group they are assigned to
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Right Motor Area Cerebellum (Experimental): Participants will receive Focused Ultrasound stimulation to motor area of the right cerebellum prior to completing a motor learning task.
  Interventions: Other: Focused Ultrasound
- Non-Motor Area Cerebellum (Experimental): Participants will receive Focused Ultrasound stimulation to a non-motor area of the right cerebellum prior to completing a motor learning task.
  Interventions: Other: Focused Ultrasound
- Control (Sham Comparator): Participants will have the Focused Ultrasound transducer placed on their neck without stimulation as a Sham present prior to completing a motor learning task.
  Interventions: Other: Sham

INTERVENTIONS:
Other: Focused Ultrasound — Low intensity focused ultrasound is sound energy stimulation at a low intensity of 1-30 W/cm2
  Arms: Non-Motor Area Cerebellum; Right Motor Area Cerebellum
Other: Sham — The investigators will simulate focused ultrasound stimulation similar to the experimental groups but without stimulation.
  Arms: Control

SUMMARY:
Transcranial focused ultrasound stimulation (tFUS) will be used in this study to functions of the cerebellum in human motor learning. Participants will complete a visuomotor task while receiving stimulation pulses from tFUS. How tFUS stimulation influencing the acquisition and retention of motor memory will be assessed based on group comparison of behavioral measures such as reaching accuracy.

DETAILED DESCRIPTION:
The purpose of this study is to test functions of the cerebellum in human motor learning. The cerebellum has been thought to play critical roles in human motor control and motor learning. Non-invasive brain stimulation studies with transcranial direct current stimulation (tDCS) and transcranial magnetic stimulation (TMS) provided evidence for the involvement of the cerebellum in human motor learning. However, due to limitations in spatial resolution of tDCS and TMS stimulation, it is still unclear what specific functions the cerebellum may have in motor learning, considering the behavioral and anatomical evidence that the cerebellum also has connections with prefrontal cortex and is associated with cognitive functions. By applying transcranial focused ultrasound stimulation (tFUS), which is a non-invasive brain stimulation technology with great spatial precision, the investigators aim to dissect functions of motor area and non-motor area of the cerebellum in motor learning. Young healthy adults will be recruited and randomly assigned to one of three experimental groups. During learning to adapt to a visual rotation (45 degrees) when reaching for a virtual target, subjects will receive tFUS stimulation over motor area of the cerebellum or non-motor area of the cerebellum depending on the study group. How tFUS stimulation influencing the acquisition and retention of motor memory will be assessed based on group comparison of behavioral measures such as reaching accuracy.

ELIGIBILITY:
Inclusion Criteria:

* Healthy, adult subjects
* 18 to 35 years of age
* Right-handed
* Provide written informed consent

Exclusion Criteria:

* Presence of a psychiatric or neurologic illness
* History of loss of consciousness of more than ten minutes in the past year or loss of consciousness in a lifetime that required rehabilitation services
* Personal or family history of seizure
* Any history of stroke/transient ischemic attack (TIA) or severe traumatic brain injury
* Taking any medications that may decrease the threshold for seizure
* Pregnancy (self-reported)
* Affirmative answers to one or more questions of the provided attached safety questionnaires. These are not absolute contraindications to this study but the risk/benefit ratio will be carefully balanced by the PI
* Have any type of metal in the body
* Failure to follow laboratory or study procedures

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 45 (Estimated)
Dates: Start 2019-01-28 (Actual); Primary Completion 2020-01-27 (Estimated); Study Completion 2020-01-27 (Estimated)

PRIMARY OUTCOMES:
Performance Error on Visuomotor Task | baseline, immediately after FUS, and 30 minutes after FUS
  The visuomotor task has practice, baseline, and experimental trials. Performance on the task will be compared between groups.

SECONDARY OUTCOMES:
Changes in Motor Evoked Potentials (MEP) | baseline, immediately after FUS, 10 minutes after FUS, and 20 minutes after FUS
  MEPs will be taken at baseline and throughout the task to assess effects ultrasound stimulation has on MEPs.

CONTACTS AND LOCATIONS:
Overall Officials: Wynn Legon, PhD, Principal Investigator — University of Virginia
Locations (1):
- University of Virginia, Charlottesville, Virginia, United States

IPD SHARING:
Plan to Share IPD: Undecided